CLINICAL TRIAL: NCT02503826
Title: The Efficacy and Optimal Dose of Sufentanil in Patient Controlled Analgesia After Moderate Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Luming Zhen, attending doctor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: LLGZB-FS-003-01
Record Dates: First submitted 2015-07-13; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Analgesia, Patient-Controlled; Gastrectomy; Arthroplasty
MeSH Terms: conditions — Agnosia | interventions — Sufentanil; Midazolam; Propofol; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- 1.5 SF (Experimental): Sufentanil,1.5mcg/kg
  Interventions: Drug: Sufentanil; Drug: Midazolam; Drug: propofol; Drug: cisatracurium
- 2.0 SF (Experimental): Sufentanil, 2.0mcg/kg
  Interventions: Drug: Sufentanil; Drug: Midazolam; Drug: propofol; Drug: cisatracurium
- 2.5 SF (Experimental): Sufentanil, 2.5mcg/kg
  Interventions: Drug: Sufentanil; Drug: Midazolam; Drug: propofol; Drug: cisatracurium

INTERVENTIONS:
Drug: Sufentanil — low dose
  Other Names: Renfu Pharmacy
  Arms: 1.5 SF
Drug: Sufentanil — moderate dose
  Other Names: Renfu Pharmacy
  Arms: 2.0 SF
Drug: Sufentanil — high dose
  Other Names: Renfu Pharmacy
  Arms: 2.5 SF
Drug: Midazolam — Midazolam 2 mg, sufentanil 0.5 mcg/kg, propofol 2 mg/kg, cisatracurium 2 mg/kg for induction, continuous infusion of propofol, remifentanil and cisatracurium to maintain bispectral index (BIS) value between 40 and 60 for maintenance.
Drug: propofol
Drug: cisatracurium

SUMMARY:
Effective postoperative pain control is essential for patients and inadequate postoperative pain relief can cause mental and psychological sufferings. Despite the growing concern on postoperative pain management, acute postoperative pain is still poorly managed. Though numerous clinical practice guidelines for postoperative pain management have been published throughout the last decades, inadequate pain relief remain a big health care issue. Sufentanil has been used as satisfied pain control drug because of its strong potency of analgesia for a long while. But its use in patient controlled intravenous analgesia (PCIA) has not been clarified. And the dilemma of safety concern and insufficient dosage of analgesic is a common problem. Thus the investigators design this prospective randomized controlled double blinded trial to observe the efficacy and the optimal dose of sufentanil in PCIA in patients underwent moderate surgery for the purpose of providing reference in clinical practice.

DETAILED DESCRIPTION:
Objective To explore the efficacy and the optimal dose of sufentanil in PCIA in patients underwent moderate surgery for the purpose of providing reference in clinical practice.

Methods 60 patients aging from 20 to 75，BMI 18 to 28 kg/m2，American Society of Anesthesiologists (ASA) grade I to II, anticipated surgery duration within 4 hrs and agreed to sign consent paper were scheduled for selective moderate surgery(including abdominal surgery and arthroplasty). Exclusive criteria: severe respiratory, cardiovascular or neurological disease, hepatic or renal dysfunction, psychiatric history or with unstable mental state, drug addiction or dependence. All patients were randomly assigned into 3 groups, S1 received 1.5 ug/kg sufentanil in PCIA, S2 received 2.0 ug/kg sufentanil, S3 received 2.5 ug/kg sufentanil. All patients received general anesthesia which was induced with midazolam 2mg, sufentanil 0.5ug/kg, propofol 2mg/kg, cisatracurium 0.2mg/kg and was maintained with continuous infusion of propofol, remifentanil and cisatracurium to maintain bispectral index (BIS) value between 40 and 60. Monitoring of MAP, heart rate (HR), pulse oxymetry (SpO2%), End-tidal CO2 (ETCO2), blood loss, and transfusion were recorded during anesthesia.

After patient waked, a loading dose of 10 ug sufentanil was given per time according to the patients' pain level and the loading dose was repeated till the pain relived or the RR was less than 10 times per min. Then the patient-controlled analgesia (PCA) pump was attached, and the continuous infusion speed was set at 2 ml/h. The pump was set to give an amount of 0.5ml at each press with a lockout interval of 10min. Patient was observed in the PACU for at least 30 min until the discharge criteria was reached. All the patients were followed-up at 2h, 6h, 24h and 48 h after the surgery. Clinical evaluations included MAP, HR, respiratory rate (RR), SpO2%, total pressing times, total amount of sufentanil, additional analgesic requirement, VAS, numerical rating scale (NRS) and Ramsey sedation scale were recorded. Side effects include nausea and vomiting, urinary retention, pruritus, respiratory depression were also recorded. Overall satisfaction index were inquired as well.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 75 years old,
* BMI 18 to 28kg/m2,
* ASA I to II grade,
* anticipated surgery duration within 4hrs,
* agree to sign consent paper.

Exclusion Criteria:

* severe respiratory,
* cardiovascular or neurological disease,
* hepatic or renal dysfunction,
* psychiatric history or with unstable mental state,
* drug addiction or dependence

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of Pain on the VAS scale after surgery | 2, 6, 24 and 48hrs after surgery
Change of Pain on the NRS scale after surgery | 2, 6, 24 and 48hrs after surgery